CLINICAL TRIAL: NCT00934050
Title: A Long-Term Follow-Up Study of Oral ELND005 (AZD-103) in Subjects With Alzheimer's Disease
Brief Title: ELND005 Long-Term Follow-up Study in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELND005-AD251
Record Dates: First submitted 2009-06-29; First posted 2009-07-08 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — scyllitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ELND005 (Experimental)
  Interventions: Drug: ELND005 (scyllo-inositol)

INTERVENTIONS:
Drug: ELND005 (scyllo-inositol) — Prior to 15Dec2009: ELND005 2000 mg PO BID for 48 weeks
  After 15Dec2009: ELND005 250 mg PO BID for 48 weeks
  Other Names: scyllo-inositol

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of ELND005 beyond the 18 months of treatment in original randomized and blinded clinical trail ELND005-AD201.

ELIGIBILITY:
Inclusion Criteria:

* This study is open only to subjects who have completed the week 78 visit in Study ELND005-AD201 while taking their assigned dose of study drug medication.

Exclusion Criteria:

* Subject has no new medical contraindications to continued participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (30):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - University of Arizona, Health Sciences Center, Dept. of Neurology, Tucson, Arizona
  - Margolin Brain Institute, Fresno, California
  - Collaborative NeuroScience Network, Inc., Garden Grove, California
  - Yale University School of Medicine, Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Brain Matters Research, Delray Beach, Florida
  - Sunrise Clinical Research, Inc, Hollywood, Florida
  - Roskamp Institute, Sarasota, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, Dept. of Neurology, Atlanta, Georgia
  - Dekalb Neurology Associates, LLC, Decatur, Georgia
  - Department of Neurology - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Department of Neurology, Kansas City, Kansas
  - Innovative Clinical Concepts, Paducah, Kentucky
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Global Medical Institutes, Princeton, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Neurological Associates of Albany, PC, Albany, New York
  - Columbia University Sergievsky Center, New York, New York
  - AD-CARE, Monroe Community Hospital, Rochester, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - Medford Neurological and Spine Clinic, Medford, Oregon
  - Summit Research Newtwork, Inc., Portland, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - University of Pittsburgh Alzheimer Disease Research Clinic, Pittsburgh, Pennsylvania
  - Butler Hospital, Memory and Aging Center, Providence, Rhode Island
  - Alliance for Neuro Research, LLC dba Absher Neurology, PA, Greenville, South Carolina
  - Clinical Neuroscience Research Associates, Inc-The Memory Clinic, Bennington, Vermont
- Canada (8):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - University of British Columbia Hospital, Division of Neurology, Vancouver, British Columbia
  - Parkwood Hospital, London, Ontario
  - Sisters of Charity of Ottawa Health Service, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Whitby Mental Health Memory Clinic, Toronto, Ontario
  - Gerontion Research, Inc., Toronto, Ontario
  - Recherche Clinique de Neurologie (Hospital Maisonneuve Rosemont), Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who enrolled in long term follow up prior to 15 Dec 2009 received ELND005 2000 mg BID; due to protocol amendment, all participants who enrolled in long term follow up after 15 Dec 2009 received ELND005 250 mg BID
Groups:
- Placebo/ELND005 2000mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive Placebo for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up prior to 15 Dec 2009 were assigned to receive ELND005 2000 mg PO BID for 48 weeks.
- 250mg/ELND005 2000mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive ELND005 250 mgPO BID for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up prior to 15 Dec 2009 were assigned to receive ELND005 2000 mg PO BID for 48 weeks.
- 1000 mg/ELND005 2000 mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive ELND005 1000 mg PO BID for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up prior to 15 Dec 2009 were assigned to receive ELND005 2000 mg PO BID for 48 weeks.
- 2000 mg ELND005/ELND005 2000 mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive ELND005 2000 mg PO BID for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up prior to 15 Dec 2009 were assigned to receive ELND005 2000 mg PO BID for 48 weeks.
- Placebo/ELND005 250 mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive Placebo for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up after 15 Dec 2009 were assigned to receive ELND005 250 mg PO BID for 48 weeks.
- 250 mg/ELND005 250 mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive ELND005 250 mg PO BID for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up after 15 Dec 2009 were assigned to receive ELND005 250 mg PO BID for 48 weeks.
Period: Enrolled Prior to 15 Dec 2009
Arm/Group | Placebo/ELND005 2000mg BID | 250mg/ELND005 2000mg BID | 1000 mg/ELND005 2000 mg BID | 2000 mg ELND005/ELND005 2000 mg BID | Placebo/ELND005 250 mg BID | 250 mg/ELND005 250 mg BID
Started | 12 | 12 | 12 | 14 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 12 | 12 | 14 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 11 | 12 | 11 | 13 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Enrolled After 15 Dec 2009
Arm/Group | Placebo/ELND005 2000mg BID | 250mg/ELND005 2000mg BID | 1000 mg/ELND005 2000 mg BID | 2000 mg ELND005/ELND005 2000 mg BID | Placebo/ELND005 250 mg BID | 250 mg/ELND005 250 mg BID
Started | 0 | 0 | 0 | 0 | 26 | 27
Completed | 0 | 0 | 0 | 0 | 19 | 23
Not Completed | 0 | 0 | 0 | 0 | 7 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo/2000mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive Placebo for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up prior to 15 Dec 2009 were assigned to receive ELND005 2000 mg PO BID for 48 weeks.
- 250mg BID/2000 mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive ELND005 250 mg PO BID for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up prior to 15 Dec 2009 were assigned to receive ELND005 2000 mg PO BID for 48 weeks.
- 1000mg BID/2000mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive ELND005 1000 mg PO BID for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up prior to 15 Dec 2009 were assigned to receive ELND005 2000 mg PO BID for 48 weeks.
- 2000mg BID/2000mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive ELND05 2000 mg PO BID for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up prior to 15 Dec 2009 were assigned to receive ELND005 2000 mg PO BID for 48 weeks.
- Placebo/ELND005 250mg BID: In the original randomized and blinded clinical trial (ELND005-AD201 NCT00568776) participants were randomized to receive Placebo for 78 weeks. Participants enrolled in ELND005-AD251 long term follow-up after 15 Dec 2009 were assigned to receive ELND005 250 mg PO BID for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo/2000mg BID | 250mg BID/2000 mg BID | 1000mg BID/2000mg BID | 2000mg BID/2000mg BID | Placebo/ELND005 250mg BID | 250 mg/ELND005 250 mg BID | Total
Number analyzed (Participants) | 12 | 12 | 12 | 14 | 26 | 27 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Enrolled prior to 15 Dec 2009 | 76.8 (5.51) | 77.0 (6.98) | 76.9 (6.92) | 69.2 (8.51) | NA (NA) — All participants enrolled after 15 Dec 2009 | NA (NA) — All participants enrolled after 15 Dec 2009 | 74.7 (7.73)
  Participants enrolled after 15 Dec 2009 | NA (NA) — All participants enrolled prior to 15 Dec 2009 | NA (NA) — All participants enrolled prior to 15 Dec 2009 | NA (NA) — All participants enrolled prior to 15 Dec 2009 | NA (NA) — All participants enrolled prior to 15 Dec 2009 | 71.4 (8.77) | 73.0 (7.53) | 72.2 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 7 | 18 | 19 | 59
  Male | 7 | 7 | 7 | 7 | 8 | 8 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 11 | 12 | 12 | 14 | 26 | 26 | 101
Region of Enrollment [Number; unit: participants]
  North America | 12 | 12 | 12 | 14 | 26 | 27 | 103

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events (TEAEs)
Description: Safety and Tolerability was assessed by the incidence of Treatment Emergent Adverse Events (TEAEs)
Time Frame: 12 months
Population: As a result of safety findings, effective 15 December 2009, all 50 patients at the 2000 mg BID dose were withdrawn from the study. Subsequently patients who were on placebo or 250 mg BID in Study AD201 received 250 mg BID in Study AD251. Only Arms who completed the study per the protocol were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo/ELND005 250mg BID | 250 mg/ELND005 250 mg BID
Number analyzed (Participants) | 26 | 27
participants | 21 | 23

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for each patient, starting from the time the consent form was signed until completion of the study (Week 54, Follow-up).
Description: For all adverse event (AE) summaries, if a patient had more than one AE within a preferred term the patient was counted once, at the maximum severity and with the closest relationship to study drug. If a patient had more than one AE within a system organ class (SOC), the patient was similarly counted once when reporting results for that SOC.
Arm/Group | Placebo/ELND005 2000mg BID | 250mg/ELND005 2000mg BID | 1000 mg/ELND005 2000 mg BID | 2000 mg ELND005/ELND005 2000 mg BID | Placebo/ELND005 250 mg BID | 250 mg/ELND005 250 mg BID
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12 | 0/12 | 2/14 | 5/26 | 6/27
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 3/14 | 11/26 | 15/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/ELND005 2000mg BID (N=12) | 250mg/ELND005 2000mg BID (N=12) | 1000 mg/ELND005 2000 mg BID (N=12) | 2000 mg ELND005/ELND005 2000 mg BID (N=14) | Placebo/ELND005 250 mg BID (N=26) | 250 mg/ELND005 250 mg BID (N=27)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Bladder transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/ELND005 2000mg BID (N=12) | 250mg/ELND005 2000mg BID (N=12) | 1000 mg/ELND005 2000 mg BID (N=12) | 2000 mg ELND005/ELND005 2000 mg BID (N=14) | Placebo/ELND005 250 mg BID (N=26) | 250 mg/ELND005 250 mg BID (N=27)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 3 | 3 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 4 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 4
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days